CLINICAL TRIAL: NCT04378075
Title: Efficacy and Safety Study of Vatiquinone for the Treatment of Mitochondrial Disease Subjects With Refractory Epilepsy
Brief Title: A Study to Evaluate Efficacy and Safety of Vatiquinone for Treating Mitochondrial Disease in Participants With Refractory Epilepsy
Acronym: MIT-E
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC743-MIT-001-EP; 2020-002100-39 (EudraCT Number)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Mitochondrial Diseases; Drug Resistant Epilepsy; Leigh Disease; Leigh Syndrome; Mitochondrial Encephalopathy (MELAS); Pontocerebellar Hypoplasia Type 6 (PCH6); Alpers Disease; Alpers Syndrome
Keywords: POLG; polymerase gamma; ALPERS; MELAS; PCH6; Pontocerebellar hypoplasia type 6; MERRF; intractable epilepsy; Mitochondrial disease; Oxidative stress; Motor seizures; Non-Motor seizures; Seizure; Refractory epilepsy; Status epilepticus; Ferroptosis; Neurodegeneration
MeSH Terms: conditions — Mitochondrial Diseases; Drug Resistant Epilepsy; Leigh Disease; Mitochondrial encephalopathy; MELAS Syndrome; Pontocerebellar Hypoplasia Type 6; Diffuse Cerebral Sclerosis of Schilder; MERRF Syndrome; Seizures; Status Epilepticus; Nerve Degeneration | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vatiquinone (Experimental): 15 milligrams/kilogram (mg/kg) if body weight <13 kg, and 200 mg if body weight ≥13 kg, administered orally, 3 times per day (TID) or up to 72 weeks
  Interventions: Drug: Vatiquinone; Other: Placebo
- Placebo (Placebo Comparator): Vatiquinone-matching placebo, administered orally, TID for up to 24 weeks followed by vatiquinone 15 mg/kg if body weight <13 kg, and 200 mg if body weight ≥13 kg, administered orally, TID for up to 48 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per the treatment arm description.
  Other Names: PTC743; EPI-743
  Arms: Vatiquinone
Other: Placebo — Vatiquinone-matching placebo will be administered per the treatment arm description

SUMMARY:
This is a parallel-arm, double-blind, placebo-controlled study with a screening phase that includes a 28-day run-in phase to establish baseline seizure frequency, followed by a 24-week, randomized, placebo-controlled phase. After completion of the randomized, placebo-controlled phase, participants may enter a 48-week, long-term, extension phase during which they will receive open-label treatment with vatiquinone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Participant or parent/legal guardian is able and willing to complete seizure diaries for the duration of the study.
* Genetic confirmation of inherited mitochondrial disease with associated epilepsy phenotype (Alpers/polymerase subunit gamma [POLG], Leigh syndrome, mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes [MELAS]), or other genetically confirmed mitochondrial disease secondary to mitochondrial mutations (Pontocerebellar Hypoplasia Type 6 [PCH6], nuclear DNA RARS2 mutation) or myoclonic epilepsy with ragged red fibers (MERRF, mitochondrial DNA [mtDNA] mitochondrially encoded tRNA lysine [MT-TK] mutation).
* Despite ongoing treatment with at least 2 antiepileptic drugs:

  * have ≥6 observed motor seizures occurring during the 28 days prior to the baseline visit (Day 0).
  * have ≥2 observed motor seizures in the first 14 days and ≥2 in the second 14 days of the Run-in period (Day -14).
  * do not have a consecutive 20-day seizure free period.
  * have at least 80% of seizure diary data.
* Documented medical history of epilepsy associated with mitochondrial disease for at least 6 months prior to screening except for participants who are <2 years of age at the time of screening (participants <2 years of age can be considered for enrollment if all other screening criteria are met due to the potential for rapid progression in these participants).
* Consent to abstain from non-approved therapies for 30 days prior to the screening visit and for the duration of the study.
* Stable dose regimen of antiepileptic therapies 30 days prior to the screening visit.
* Stable regimen of dietary supplements 30 days prior and, if on a ketogenic diet, stable ketogenic diet 90 days prior to the screening visit and for duration of the study.
* Electroencephalogram (EEG) at screening or historical EEG up to 6 months prior to screening for diagnostic confirmation of seizures.

Exclusion Criteria:

* Allergy to vatiquinone or sesame oil.
* Aspartate transaminase (AST) or alanine transaminase (ALT) ≥3 × upper level of normal (ULN) at time of screening.
* International normalized ratio (INR) >ULN at time of screening.
* Serum creatinine ≥1.5 × ULN at time of screening.
* Participation in another interventional clinical trial 60 days prior to randomization or for the duration of this clinical trial
* Previously received vatiquinone.
* Concomitant treatment with drug(s) that have not received regulatory agency approval for the treatment of mitochondrial diseases and use of artisanal (non-Epidiolex cannabidiol) cannabidiol therapies.
* Concomitant treatment with idebenone.
* Ongoing treatment with strong cytochrome P450 (CYP) inhibitors such as itraconazole or strong CYP inducers such as rifampin. Treatment with these agents must be completed at least 4 weeks prior to enrollment.During the study, participants should not use grapefruit/grapefruit juice or St John's wort extract.
* Pregnant or lactating participants or those male or female sexually active participants who are unwilling to comply with proper birth control methods from the time consent is signed until 30 days after treatment discontinuation. Females of childbearing potential must have a negative pregnancy test at screening and during the baseline visit (Day 0).
* Comorbidities that may confound study results (for example, fat malabsorption syndrome, other mitochondrial disorders) in the opinion of the investigator.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline to Week 24 in the Number of Observable Motor Seizures per 28 Days | Day 0, Week 24

SECONDARY OUTCOMES:
Number of Disease-Related Hospital Days | Week 24 and up to Week 72
Number of Participants with Occurrences or Recurrence of Status Epilepticus | Week 24 and up to Week 72
Number of Participants with Disease-Related In-Patient Hospitalizations or Emergency Room Visits | Week 24 and up to Week 72
Number of Disease-Related In-Patient Hospital Admissions or Emergency Room Visits | Week 24 and up to Week 72
Percent Change From Baseline to Week 72 in Total Seizure Frequency per 28 Days | Day 0, Week 24, Week 72
Percentage of Participants with ≥25%, ≥50%, ≥75%, and 100% Reduction in Motor Seizures | Week 24 and up to Week 72
Percentage of Participants with ≥25%, ≥50%, ≥75%, and 100% Reduction in Total Seizures | Week 24 and up to Week 72
Number of Participants Who Require Rescue Seizure Medication | Week 24 and up to Week 72
Health-Related Quality of Life as Measured by the Care-Related Quality of Life of Informal Caregivers (CarerQoL-7D) Questionnaire | Week 24 and up to Week 72
Number of Participants with Seizure Clusters | Week 24 and up to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Penematsa, MD, Study Director — PTC Therapeutics
Locations (27):
- United States (12):
  - University of California, San Diego, California
  - Stanford University, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Children's National Medical Center - Department Of Neurology, Washington D.C., District of Columbia
  - John Hopkins Medicine, Baltimore, Maryland
  - Pediatric Genetics Clinic (Main MGH Hospital), Boston, Massachusetts
  - Boston Children Hospital, Boston, Massachusetts
  - Children's of Minnesota, Minneapolis, Minnesota
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science, Houston, Texas
  - Seattle Children's hospital, Seattle, Washington
- Alberta Children's Hospital, University of Calgary, Calgary, Canada
- France (4):
  - CHU d'Angers - Service de génétique, Angers
  - CHU de Montpellier - Hôpital Gui de Chauliac - Département de neuropédiatrie, Montpellier
  - A.P.H.P - Hôpital Necker-Enfants Malades - Service de Neurologie pédiatrique, Paris
  - CHU de Strasbourg - Hôpital de Hautepierre - Service de Neuropédiatrie, Strasbourg
- Italy (2):
  - UOC Neuropsichiatria Infantile, Istituto Neurologico Carlo Besta-Fondazione IRCCS, Milan
  - U.O.C. Malattie Muscolari e Neurodegenerative, Dipartimento di Scienze Neurologiche e Psichiatriche, Ospedale Pediatrico Bambino Gesù, Roma
- PTC Clinical Site, Multiple Locations, Japan
- Instytut Pomnik-Centrum Zdrowia Dziecka, Centrum Wsparacia Pediatrycznych Badań Klinicznych, Warsaw, Poland
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Ruber Internacional, Neurology Department, Epilepsy Program, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Karolinska University hospital, Astrid Lindgrens Children Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided